CLINICAL TRIAL: NCT02164149
Title: Length of Tumour Feeding Artery After Colon Cancer Surgery
Acronym: ColonCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: CT121177
Record Dates: First submitted 2014-06-02; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Colon Cancer
Keywords: Colon cancer; Quality of surgery; Length of tumour feeding artery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quality of colon cancer surgery: Patients with primary colon cancer
  Interventions: Other: Patients with primary colon cancer

INTERVENTIONS:
Other: Patients with primary colon cancer — CT scan two days after surgery

SUMMARY:
The quality of colon cancer surgery is highly debated these years since the mortality of the disease is not declining markedly. Surgery is the main treatment of colon cancer and during surgery it is very important for the surgeon to remove the tumour and all potential ways of tumour spread. As colon cancer first of all spreads to the nearby lymph nodes lying along the tumour feeding artery the surgeon aims to cut the vessel as central as possible. This means that all of the tumour feeding artery should have been removed after surgery.

In this study the investigators want to measure the length of the tumour feeding artery after surgery as a quality control of the surgery. The investigators hypothesize that the artery will be shorter than 5 mm.

The investigators wish to CT scan all patients two days after colon cancer surgery and afterwards measure then length of the artery on the images. This study will not inflict with the normal routine for patient information and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Primary colon cancer

Exclusion Criteria:

* Kidney failure, allergy to contrast, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years with primary colon cancer, who are to have surgery at Randers Regional Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
CT scan after colon cancer surgery. The length of the tumour feeding artery will be measured on the images. | 6 to 9 months
  Patients will have an extra CT scan two days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Soren Laurberg, Professor, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark